CLINICAL TRIAL: NCT06395220
Title: Kinectics of Donor-specific Anti-HLA Antibody After HLA-incompatible Allogeneic Haematopoietic Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); Peking University First Hospital (Other); The First Hospital of Jilin University (Other); First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Chang Yingjun, Professor and Chief Physician, Peking University
Other Study IDs: PekingUPH Chang Yingjun
Record Dates: First submitted 2024-04-24; First posted 2024-05-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Haematological Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Detection of donor-specific anti-HLA antibody (DSA) — Detection methods
  1. . Morphology: using microscope to observe the morphology of bone marrow.
  2. . Immunophenotyping: using multi-color flow cytometry (MFC) to detect immunophenotype of leukemia cells and leukemia-associated immunophenotype of bone marrow samples.
  3. . Cytogenetics analysis: G-band and/or fluorescence in situ hybridization (FISH) analysis are used in this study
  4. . Molecular detection: Real-time quantitative RT-PCR (RQ-PCR) and/or next generation sequencing techniques are used to detect the molecular marker, such as: PML/RARA, AML-ETO, BCR/ABL, and WT1.
  5. . HLA-Typing: HLA-A, -B, -C, -DRB1, -DQB1, and -DPB1 alleles were determined according to the literatures published by our group [Huo MR, et al. Bone Marrow Transplant. 2018;53(5):600-608]..
  6. . Other analyses: Detection of minimal residual diseases were performed using MFC and RQ-PCR according to the methods reported by our group [Li SQ, et al. Blood,2022;140(5):516-520].

SUMMARY:
Donor specific anti-HLA antibody (DSA) is closely related not only to primary graft rejection (GR) after HLA-incompatible transplantation, but also to the occurrence of primary PGF. Desensitisation therapy can reduce the level of DSA in patients and decrease the incidence of PGF after transplantation. However, most studies at home and abroad have focused on DSA levels in recipients before transplantation, risk factors and their effects on prognosis. Very few studies have focused on the rate of DSA positivity and its risk factors after transplantation. Therefore, this project aims to clarify the rate of DSA positivity after HLA-incompatible Allo-HSCT and reveal the influencing factors of post-transplantation DSA positivity with the help of a prospective, registry-based clinical cohort of HLA-incompatible transplant recipients, in order to provide a basis for the prevention and treatment of DSA-induced graft rejection or PGF.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis haematological disorders undergoing HLA-incompatible allogeneic haematopoietic stem cell transplantation Between 15 and 60 years-old Must sign the informed consent

Exclusion Criteria:

Withdraw of the signed informed consent for any reason Lack of ability to provide consent due to psychiatric or physical illness

Ages: 15 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: The basis of sample selection of 800 cases, according to the data of our centre, pre-transplant DSA-positive patients accounted for 11.3% of all transplanted patients, DSA-positive patients given desensitisation treatment before transplantation had a DSA-positive rate of 7% after transplantation, and 710 pre-transplant DSA-negative patients had a post-transplant DSA-positive rate of 7%, so it was 50 cases, and the total number of DSA-positive cases was 56 cases; The above calculations were made without desensitisation of pre-transplant DSA-positive patients and the post-transplant DSA-positive rate of pre-transplant DSA-negative patients was calculated according to pre-transplant DSA-positive patients.
Sampling Method: Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Positive rates of post-transplantation donor-specific anti-HLA antibody (DSA). | through study completion, an average of 2 years
  HLA-A, -B, -C, -DRB1, -DQB1, and -DPB1 alleles were determined according to the literatures published by our group [Huo MR, et al. Bone Marrow Transplant. 2018;53(5):600-608].

SECONDARY OUTCOMES:
Acute graft-versus-host disease (aGVHD) | 2 years
  Acute GVHD was defined and graded from I to IV based on the pattern and severity of organ involvement [Sullivan KM. Graft-versus-host-disease. In: Thomas ED, Blume KG, Forman SJ (eds). Hematopoietic Cell Transplantation. 5nd edn. Blackwell Science: Boston, MA, USA, 2020, pp 515-536.].
Chronic graft-versus-host disease (cGVHD) | 2 years
  Chronic GVHD was defined and graded according to the National Institute of Health criteria:[Biol Blood Marrow Transplant,2005,11: 945] that is, mild cGVHD reflects the involvement of no more than 1 or 2 organs/sites (except for lung) with a maximum score of 1; moderate cGVHD involves at least 1 organ/site with a score of 2 or ≥3 organs/sites with a score of 1 (or lung score 1); and severe cGVHD is diagnosed when a score of 3 is given to any organ (or lung score 2). The diagnosis is mainly based on clinical manifestations.
Neutrophil engraftment | 2 years
  Neutrophil engraftment was defined as the first day of an absolute neutrophil count above 0.5×109/L for three consecutive days after the neutrophil nadir.
Platelet engraftment | 2 years
  Platelet engraftment was defined as the first of 7 consecutive days during which the platelet count was at least 20×109/L without needing transfusion.
Primary graft failure | 2 years
  Primary graft failure was defined as never achieved an ANC >0.5×109/L for thress consecutive days or an ANC >0.5×109/L without donor engraftment (autologous recovery).
Secondary graft-failurefunction | 2 years
  Secondary graft-failure was defined as decline or loss of donor engraftment.
Cumulative incidence of relapse | 2 years
  Relapse was defined by the morphological evidence of disease in the peripheral blood, BM or extramedullary sites. Time to relapse was defined from the date of transplantation to the date of disease recurrence. Patients exhibiting minimal residual disease (for example, the presence of BCR/ABL RNA transcripts by PCR) were not classified as having morphological relapse.
Non-relaspe mortality (NRM) | 2 years
  Non-relapse mortality was defined as all causes of death other than those related directly to malignant disease itself, occurring at any time after transplantation.
Disease-free survival (LFS) | 2 years
  Disease-free survival was defined as days from transplantation to disease progression after transplantation.
Overall survival (OS) | 2 years
  Overall survival referred to patients who survived until the final follow-up time point.

CONTACTS AND LOCATIONS:
Locations (1):
- People's Hospital of Peking University, Beijing, China

IPD SHARING:
Plan to Share IPD: No